CLINICAL TRIAL: NCT04307485
Title: A Randomized Controlled sTudy of Low Dose vs Standard tIcaGrelor on Platelet Function After intErvention for Acute Coronary syndRome in Senior Patients
Brief Title: A Study of Low Dose vs Standard Ticagrelor on Platelet Function After Intervention for Acute Coronary Syndrome in Senior Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Principal Investigator, Hou Lei, Clinical Professor, Shanghai Tong Ren Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020HL
Record Dates: First submitted 2020-03-08; First posted 2020-03-13 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Senior Acute Coronary Syndrome Patients After PCI
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard dose ticargrelor based DAPT therapy (Active Comparator): treated with ticagrelor 90mg and aspirin 100mg after PCI for 12 months as the standard group
  Interventions: Drug: Ticagrelor
- low dose ticargrelor based DAPT (Experimental): treated with ticagrelor 60mg plus aspirin 100 mg for 11 months after one month standard DAPT treatment
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — 90mg ticargrelor based DAPT vs 60mg ticargrelor based DAPT

SUMMARY:
In this study, the investigates try to confirm our hypothesis that low dose ticagrelor(60mg) had similar anti-platelets function compared with the standard dose ticagrelor in senior （no less than 75 years old)acute coronary syndrome patients . Totally 40 senior ACS patients will be divided into 2 groups randomly one month after PCI . Group 1 will be treated with ticagrelor 90mg and aspirin 100mg after PCI for 12 months as the standard group; Group 2 will be treated with ticagrelor 60mg plus aspirin 100 mg for 11 months after one month standard DAPT treatment. The platelets function will be tested in VASP and TEG methods 2 months after PCI as the primary endpoints.The clinical events will be observed 12 months after PCI.

ELIGIBILITY:
Inclusion Criteria:

1.Subject must be at least 75 years of age 2 Patients should have undergone successful percutaneous coronary intervention with drug-eluting stent for acute coronary syndrome 3.Subject understand the study requirements and the treatment procedures and provided informed consent before the procedure

Exclusion Criteria:

1. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
2. Active bleeding
3. Known hypersensitivity or contraindication to study medications
4. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
5. Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment).
6. Subjects with Cerebral hemorrhage history
7. Subjects with stroke history in half a year
8. subjects with active malignant tumor
9. subjects with whom oral anticoagulants are needed
10. Other conditions which the investigators think not applicable to the study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
changes of PRI detected by VASP methods | changes of PRI from baseline (4weeks after index PCI) to 8 and 12 weeks after index PCI
  platelet reactivity index (PRI) detected by VASP (Vasodilator Stimulated
changes of Maximum Amplitude (MA) detected by TEG | changes of MA from baseline (4weeks after index PCI) to 8 and 12 weeks after index PCI
  Maximum Amplitude (MA) detected by TEG(Thromboelastography)

CONTACTS AND LOCATIONS:
Locations (1):
- shanghai Tongren hospital, Shanghai, Shanghai Municipality, China